CLINICAL TRIAL: NCT06307054
Title: The Safety and Efficacy for Anti-human CLL-1 CAR-NK Cells in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: CLL-1 CAR-NK Cells for Relapsed/Refractory AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Doctor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSY-CAR-NK-AML01
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Adult AML; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti CLL-1 CAR NK cells (Experimental)
  Interventions: Drug: anti-CLL-1 CAR NK cells

INTERVENTIONS:
Drug: anti-CLL-1 CAR NK cells — Eligible patients enrolled in the study after screening will receive lymphocyte collection(from the patient or a donor ) and receive single dose CLL-1 CAR NK cells infusion after a successful cell production. There are a total of four cell dose level:5×10^6 CAR-NK cells/kg,1×10^7CAR-NK cells/kg,2×10^7CAR-NK cells/kg,4×10^7CAR-NK cells/kg

SUMMARY:
This study is a single-arm, open-label, dose-escalation clinical trial aimed at exploring the safety, tolerability, and pharmacokinetic characteristics of the CLL-1 CAR NK cells, as well as providing preliminary observations on its efficacy in subjects with relapsed/refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years, gender unrestricted;
2. Expected survival time exceeds 12 weeks;
3. ECOG score 0-2;
4. Meets the 2022 WHO criteria for acute myeloid leukemia and flow cytometry shows ≥70% expression of CLL1 in leukemia cells; or immunohistochemistry shows CLL1 expression ≥50% and meets the following criteria for relapse and refractory:

   1. Relapse criteria: Bone marrow shows primitive cells ≥5% after hematological remission (excluding post-chemotherapy hematopoietic recovery); or at least two peripheral blood samples taken at least one week apart show primitive cells; or extramedullary lesions are present. Early relapse (relapse within 12 months after initial remission) patients can be directly included, while late relapse (relapse after 12 months of initial remission) patients must have undergone salvage chemotherapy according to standard protocols without achieving complete remission. Salvage treatment for all relapsed patients should include at least one course of targeted therapy without achieving remission. Patients who relapse after allogeneic hematopoietic stem cell transplantation, have no other effective treatment options, and have no active grade 2 or higher acute GVHD.
   2. Refractory criteria: No complete remission after two courses of standard intensive chemotherapy based on the 3+7 regimen, and no complete remission after second-line salvage chemotherapy or treatment including targeted therapy; or no complete remission after one course of purine analog induction chemotherapy (such as FLAG-Ida, CLIA, or similar regimens), and no complete remission after salvage treatment or treatment including targeted therapy; or no complete remission after three cycles of low-intensity treatment based on HMA, including low-intensity regimens containing venetoclax; relapse within 12 months after remission (early relapse); patients for whom the original induction is ineffective after relapse.
5. Able to establish the required venous access for collection, and no contraindications for leukapheresis;
6. Liver and kidney function, cardiac and pulmonary function meet the following requirements:

   1. Creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 60 mL/min or creatinine ≤ 2.5×ULN;
   2. Ejection fraction >50%, no clinically significant electrocardiogram changes; baseline blood oxygen saturation >92%; total bilirubin ≤ 3×ULN; ALT and AST ≤ 3×ULN;
7. Able to understand and sign the informed consent form.

Exclusion Criteria:

Any of the following conditions disqualify a subject from participation in the trial:

1. Confirmed AML with PML-RARA fusion gene;
2. History of malignancies other than acute myeloid leukemia within 5 years before screening, except adequately treated carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin, or prostate cancer after radical surgery, or thyroid cancer after radical surgery;
3. Uncontrolled active bacterial, viral, or fungal infections requiring treatment; HBsAg or HBcAb positive, with peripheral blood HBV DNA ≥ lower limit of detection; HCV RNA positive in the presence of hepatitis C virus antibodies; positive TRUST test for syphilis; HIV antibody positive;
4. Significant organ (cardiovascular, pulmonary) dysfunction; active gastrointestinal bleeding within the past 3 months; uncontrolled hypertension or history of hypertensive crisis or hypertensive encephalopathy; significant history or evidence of major cardiovascular risk, including congestive heart failure, unstable angina, clinically significant arrhythmias (such as ventricular fibrillation, ventricular tachycardia, etc.); history of arterial thrombosis within the past 3 months (such as stroke, transient ischemic attack); symptomatic deep vein thrombosis within the past 6 months, history of pulmonary embolism, or history of coronary angioplasty, defibrillation, or any clinical significant complications or diseases that may pose a risk to the subject's safety or interfere with the study evaluation, procedures, or completion;
5. Any uncontrolled active disease that hinders participation in the trial;
6. Active, uncontrolled central nervous system involvement, or a history of central nervous system disease requiring treatment (such as epilepsy);
7. Subjects receiving systemic corticosteroid therapy before screening and deemed by the investigator to require long-term systemic corticosteroid therapy during the study period (excluding inhalation or local use); and subjects who have received systemic corticosteroid therapy within 72 hours before cell infusion (excluding inhalation or local use);
8. Subjects who have used PD-1 or PD-L1 monoclonal antibodies within 3 months before enrollment
9. Pregnant or lactating women; and subjects planning to become pregnant within 1 year after infusion, during or after the treatment period;
10. Uncontrolled active infections (excluding simple urinary tract infections or upper respiratory tract infections);
11. Subjects who have received CAR-T therapy or other gene-modified cell therapy in the past;
12. Patients after allogeneic transplantation, with no significant acute or chronic GVHD, and have discontinued immunosuppressive drugs for at least 1 month;
13. Known allergy to any component of anti-CLL-1 CAR-NK cell infusion or chemotherapy regimen (cyclophosphamide and fludarabine);
14. Any situation deemed by the investigator to compromise the safety of the subject or interfere with the purpose of the study, or deemed unsuitable for participation by the investigator;
15. Afflicted with a condition that affects the ability to sign the informed consent form in writing or to comply with the study procedures; unwilling or unable to comply with the study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
AE | 14 days-28 days after infusion
  Adverse events related to cell reinfusion (≥ Grade 3 treatment-related organ toxicity, laboratory tests, and Grade 4 hematologic toxicity, etc.);
DLT | 14 days-28 days after infusion
  Dose limited toxicity

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 28 days after infusion
  PK parameters: the maximum concentration (Cmax) of anti-CLL-1 CAR-NK cells in peripheral blood after administration, time to reach maximum concentration (Tmax), and area under the curve
PD | Time points according to the study
  PD parameters: content of T/NK cells in peripheral blood (detection includes CD3, CD4, CD7, CD8, CD16, CD56, CD25, FOXP3, etc.); plasma cytokine levels at various time points;
Complete response | 28 days after infusion
  Complete response
Duration of response (DOR) | 28 days after infusion
  the time from the first assessment of CR or CRi or PR to the first assessment of disease progression or death for any reason
Progression-free survival (PFS) | through study completion, an average of 2 years
  the time from cell reinfusion to the first assessment of tumor progression, relapse, or death for any reason
Overall survival (OS) | through study completion, an average of 2 years
  the time from cell reinfusion to death for any reason
Number of participants with treatment-related AEs as assessed by CTCAE v5.0 | through study completion, an average of 2 years
  Liver and kidney function

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No